CLINICAL TRIAL: NCT02585245
Title: Comparison of Nutrition Risk Screens in Identification of Hospitalized Patients at Nutrition Risk and/or With Malnutrition.
Brief Title: Comparison of Nutrition Risk Screens
Status: Completed | Type: Observational
Sponsor: ThedaCare (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: TC0001
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2016-10

CONDITIONS: Malnutrition
Keywords: Hospital Nutrition screens
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NRS2002 Nutrition Risk Screen: Patients identified at HIgh, medium or Low Risk in Hospitalized patients. Determining accuracy of identifiying patients affected by malnutrition.
- ThedaCare RD/RN Nutrition Risk Screen: Patients identified at HIgh, medium or Low Risk in Hospitalized patients. Determining accuracy of identifiying patients affected by malnutrition.

SUMMARY:
This research study will compare two different screens for nutrition risk in patients who are in the hospital. We will be comparing the ThedaCare Nutrition Risk Screen to see if it is as good and consistent as the standard NRS 2002 Nutrition Risk Screen.

DETAILED DESCRIPTION:
This research study comparing the ThedaCare screen against the NRS 2002 screen will validate the accuracy and reliability of the ThedaCare Screen and the timeliness of nutrition intervention of patients with a diagnosis of malnutrition. Early nutrition intervention will positively affect the patient's clinical complication, LOS, and readmission.

ELIGIBILITY:
Inclusion Criteria:

* 18 yrs of age
* Hopitalized

Exclusion Criteria:

* Positve for Pregnancy
* Inability to give Consent

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Hospitalized patients that can consent
Sampling Method: Non-Probability Sample
Enrollment: 607 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori LK Hartz, MS, RDN, Principal Investigator — ThedaCare
Locations (2):
- United States (2):
  - ThedaCare Regional Medical Center- Appleton, Appleton, Wisconsin
  - ThedaCare Regional Medical Center, Neenah, Wisconsin

REFERENCES:
- [Background] Malone A, Hamilton C. The Academy of Nutrition and Dietetics/the American Society for Parenteral and Enteral Nutrition consensus malnutrition characteristics: application in practice. Nutr Clin Pract. 2013 Dec;28(6):639-50. doi: 10.1177/0884533613508435. Epub 2013 Oct 31. PMID 24177285
- [Background] Kyle UG, Kossovsky MP, Karsegard VL, Pichard C. Comparison of tools for nutritional assessment and screening at hospital admission: a population study. Clin Nutr. 2006 Jun;25(3):409-17. doi: 10.1016/j.clnu.2005.11.001. Epub 2005 Dec 13. PMID 16356595
- [Background] Kondrup J, Allison SP, Elia M, Vellas B, Plauth M; Educational and Clinical Practice Committee, European Society of Parenteral and Enteral Nutrition (ESPEN). ESPEN guidelines for nutrition screening 2002. Clin Nutr. 2003 Aug;22(4):415-21. doi: 10.1016/s0261-5614(03)00098-0. PMID 12880610
- [Background] Corkins MR, Guenter P, DiMaria-Ghalili RA, Jensen GL, Malone A, Miller S, Patel V, Plogsted S, Resnick HE; American Society for Parenteral and Enteral Nutrition. Malnutrition diagnoses in hospitalized patients: United States, 2010. JPEN J Parenter Enteral Nutr. 2014 Feb;38(2):186-95. doi: 10.1177/0148607113512154. Epub 2013 Nov 18. PMID 24247093
- [Background] Makhija S, Baker J. The Subjective Global Assessment: a review of its use in clinical practice. Nutr Clin Pract. 2008 Aug-Sep;23(4):405-9. doi: 10.1177/0884533608321214. PMID 18682592
- [Derived] Hartz LLK, Stroup BM, Bibelnieks TA, Shockey C, Ney DM. ThedaCare Nutrition Risk Screen Improves the Identification of Non-Intensive Care Unit Patients at Risk for Malnutrition Compared With the Nutrition Risk Screen 2002. JPEN J Parenter Enteral Nutr. 2019 Jan;43(1):70-80. doi: 10.1002/jpen.1315. Epub 2018 Jun 30. PMID 29959847

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All patients received both the NRS 2002 and the ThedaCare Nutrition Risk Screen. Patients identified at HIgh, medium or Low Risk in Hospitalized patients. Determining accuracy of identifiying patients affected by malnutrition.
Period: Overall Study
Arm/Group | All Participants
Started | 607
Completed | 594
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 594
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 318
  Male | 276
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 594

OUTCOME MEASURES:

1. Primary Outcome: The Percent of Participants Identified With Malnutrition Using the NRS 2002 and ThedaCare Nutrition Risk Screen
Description: Sensitivity: True Positives/ (True Positives +False Negatives) Specificity: True Negatives/ (True Negatives + False Positives)
Time Frame: 24 hr within admission to the hospital
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NRS2002 Nutrition Risk Screen | ThedaCare RD/RN Nutrition Risk Screen
Number analyzed (Participants) | 594 | 594
percentage of participants
  Sensitivity | 63.5 [58.3 to 68.7] | 98.8 [97.6 to 99.9]
  Specificity | 94.3 [91.5 to 97.1] | 74 [68.7 to 79.2]

ADVERSE EVENTS:
Description: Adverse events were not assessed.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 113/594
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes